CLINICAL TRIAL: NCT01263054
Title: A Prospective, Randomized, Multi-Center, Open-Label Clinical Trial Comparing Disc Biacuplasty With Medical Management for Discogenic Lumbar Back Pain
Brief Title: Safety and Efficacy of the TransDiscal System Versus Medical Management in Treating Chronic Discogenic Low Back Pain
Acronym: COLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halyard Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100-10-0001
Record Dates: First submitted 2010-11-29; First posted 2010-12-20 (Estimated); Results first posted 2016-03-09 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2015-03

CONDITIONS: Back Pain
Keywords: Back Pain; Low Back Pain; Discogenic Back Pain
MeSH Terms: conditions — Back Pain; Low Back Pain | interventions — Practice Management, Medical; Physical Therapy Modalities; Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TransDiscal System (Experimental): Kimberly-Clark TransDiscal System in addition to standard medical management
  Interventions: Device: TransDiscal System
- Medical Management (Other): Standard medical management
  Interventions: Other: Medical Management

INTERVENTIONS:
Device: TransDiscal System — Surgical Procedure using the TransDiscal System to perform disc biacuplasty.
  Other Names: TransDiscal,disc biacuplasty,disc,ablation,low back pain
  Arms: TransDiscal System
Other: Medical Management — Standard medical management, physical therapy, and lifestyle changes.
  Other Names: physical therapy, medications,
  Arms: Medical Management

SUMMARY:
The primary objective of this randomized controlled trial is to evaluate the safety and efficacy of the TransDiscal System (TDS) in treating discogenic pain of the lumbar spine using a modified disc biacuplasty procedure. The primary efficacy measure will be the Visual Analog Scale (VAS) at 6 months post treatment/randomization and the TransDiscal System will be compared against medical management (standard of care).

DETAILED DESCRIPTION:
The intervertebral discs serve as joints between the vertebral bodies, providing both structural support and flexibility to the spinal column. Intervertebral discs do not remain structurally intact over a lifetime and degenerate as a natural part of aging. Degenerated discs do not react to stresses and forces the same as healthy discs. When too much stress is applied to a degenerated disc, tears can result. Evidence suggests that when a tear is present, sensory nerve endings can grow into the tear and transmit pain.

The TransDiscal System (TDS) is a medical device that is used in a procedure called Disc Biacuplasty and is currently available in the United States and throughout the world. The TDS enables the back of the disc to be heated to high enough temperatures to ablate the nerves inside that are transmitting pain, while maintaining low enough temperatures to prevent damage to surrounding tissues. The TDS uses two electrodes, located at the ends of two thin probes, which are placed on both sides of the back of the intervertebral disc by inserting them through the skin into the disc using x-ray guidance. Radiofrequency (RF) current flows in the disc between the two electrodes, heating the tissue in the disc to the desired temperature. The study evaluates a modified heating protocol than what is currently in clinical use which should allow for a larger area of the back of the disc to be heated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥21 years
* Able to understand the informed consent and able to complete outcome measures
* Objective measurements indicating functional impairment related to low back pain
* Stabilized on pain medication regimen for >2 months as defined by a <10% change in dosage
* History of chronic low back pain (>6 months) unresponsive to non-operative care (including physical therapy, anti-inflammatory medication, epidurals, diagnostic facet joint/medial branch blocks, and sacroiliac joint interventions as performed or deemed appropriate by the Investigator)
* Score ≥5 on the Visual Analog Scale (VAS) relating specifically to the average daily low back pain
* Back pain more prominent than leg pain which is commonly exacerbated by flexion or bending or prolonged sitting.
* Single level concordant pain reproduction present on lumbar discography in desiccated disc. Magnetic resonance Imaging (MRI) image also supports discography findings. Changes in other disc spaces in the lumbar region do not demonstrate neural compressive lesion.
* Disc height at least 50% of adjacent control disc

Exclusion Criteria:

* Evidence of compressive radiculopathy with predominant leg pain
* Evidence of nucleus pulposus herniation or free disc fragments on MRI
* Evidence of > 2 discs dessicated based on MRI or symptomatic involvement of more than one lumbar disc levels.
* Asymptomatic disc bulges > 5 mm at the treatment level.
* Prior lumbar surgery of any kind at the treatment level (micro-discectomies, and/or minimally invasive procedures at other levels that are not excluded)
* Prior spinal fusion below the T10 Level
* Symptoms or signs of lumbar canal stenosis at any level
* Evidence of structural abnormality at the lumbar level (except non-symptomatic spondylolysis resulting in spondylolithesis no more than Grade 1 upon flexion and extension)
* Any generalized pain or multifocal pain,conversion or multiple non-anatomical complaints
* Pending or active compensation claim, litigation or disability income remuneration (secondary gain)
* Chronic pain associated with significant psychosocial dysfunction
* Beck's Depression Index (BDI) score >20
* Current pregnancy, recent delivery (within 3 months of consent) or the intent of becoming pregnant during the study period.
* Systemic or localized infection at the anticipated needle entry site (subject may be considered for inclusion once infection is resolved)
* Discitis
* Allergies to any medication to be used in the procedure
* Present symptomatic lumbar spinal fracture
* History of uncontrolled coagulopathy, ongoing coagulation treatment or unexplained or uncontrollable bleeding that is uncorrectable
* Progressive neurological deficits
* Within the preceding 2 years, subject has suffered from active narcotic addiction, substance abuse or alcohol abuse
* Current prescribed opioid medications equivalent to >120 mg of morphine per 24 hours
* Uncontrolled immunosuppression (e.g. Acquired Immune Deficiency Syndrome [AIDS], cancer, diabetes, etc.)
* Body Mass Index (BMI) >32.5 kg/m^2
* Participating in another clinical trial/investigation 30 days prior to signing informed consent
* Negative or indeterminate lumbar discography results as assessed per International Spine Intervention Society (ISIS) guidelines
* Subject unwilling or unable to comply with follow up schedule or protocol requirements.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2010-12; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Curd, MS, Study Director — Halyard Health, Inc.
Locations (9):
- United States (9):
  - George Washington University Hospital, Washington D.C., District of Columbia
  - Compass Research, Orlando, Florida
  - Millennium Pain Center, Bloomington, Illinois
  - Metro Orthopedics & Sports Therapy, Silver Spring, Maryland
  - PainCare, Linwood, New Jersey
  - Center for Clinical Research, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - JPS Orthopedic & Sports Medicine, Arlington, Texas
  - Center for Pain Relief, University of Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this study, 67 subjects were randomized, with 63/67 being treated. Three of the non-treated subjects had exclusion criteria violations, while the fourth subject was not treated for an undisclosed reason. The disposition of subjects in the Participant Flow summary is with respect to the primary outcome.
Period: Overall Study
Arm/Group | TransDiscal System | Medical Management
Started | 29 | 34
Completed | 24 | 28
Not Completed | 5 | 6
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Qualification Violation | 1 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TransDiscal System | Medical Management | Total
Number analyzed (Participants) | 29 | 34 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 34 | 62
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (11) | 43 (11) | 42 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 13 | 15 | 28
Region of Enrollment [Number; unit: participants]
  United States | 29 | 34 | 63

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Daily Pain Visual Analog Scale (VAS) Score Between Screening and Follow up.
Description: Visual Analog Scale (NRS) - score range = 0 - 10. "0" corresponds to "no pain" and "10" indicates "worst pain imaginable". The means of these scores and their respective standard deviations are reported for each study group.
Time Frame: Baseline and 6 months
Population: Five subjects in the TransDiscal System study arm, and six subjects in the Medical Management study arm did not provide follow-up data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TransDiscal System | Medical Management
Number analyzed (Participants) | 24 | 28
units on a scale | -2.4 (2.8) | -0.56 (1.6)

2. Secondary Outcome: Percentage of Study Group Subjects With Greater Than 2 Points Decrease or 30% Drop in Average Daily Pain Related Visual Analog Scale (VAS) Score.
Description: as for outcome 1
Time Frame: Baseline and 6 months
Measure: Number; unit: percentage of study group
Arm/Group | TransDiscal System | Medical Management
Number analyzed (Participants) | 29 | 34
percentage of study group | 50 | 18

3. Secondary Outcome: Mean Change in Score of Short Form 36-Physical Functioning (SF36-PF) From Screening to 6 Month Follow up Visit
Description: Short Form 36-PF - score range = 0 - 100. "0" corresponds to "greatest disability" and "100" indicates "no disability". The means of these scores and their respective standard deviations are reported for each study group.
Time Frame: Baseline and 6 months
Population: Five subjects in the TransDiscal System study arm, and seven subjects in the Medical Management study arm did not provide follow-up data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TransDiscal System | Medical Management
Number analyzed (Participants) | 24 | 27
units on a scale | 18 (23) | 1.7 (16)

4. Secondary Outcome: Mean Change in Score of EuroQuol 5d Visual Analog Scale (EQ-5d VAS) Between Screening and 6 Month Follow up Visit
Description: EQ-5d VAS - score range = 0 - 100. "0" corresponds to the "worst imaginable health state" and "100" indicates the "best imaginable health state". The means of these scores and their respective standard deviations are reported for each study group.
Time Frame: Baseline and 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TransDiscal System | Medical Management
Number analyzed (Participants) | 24 | 27
units on a scale | 15 (42) | 6 (31)

5. Secondary Outcome: Mean Change in Score of Beck's Depression Inventory (BDI) Between Screening and 6 Month Follow up Visit
Description: BDI - score range = 0 - 63. "0" corresponds to "minimal depression" and "63" indicates "severe depression". The means of these scores and their respective standard deviations are reported for each study group.
Time Frame: Baseline and 6 months
Population: Five subjects in the TransDiscal System study arm, and eight subjects in the Medical Management study arm did not provide follow-up data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TransDiscal System | Medical Management
Number analyzed (Participants) | 24 | 26
units on a scale | 0.39 (8) | -0.23 (4)

6. Secondary Outcome: Mean Change in Score of Patient Global Impression of Change (PGIC) Between Screening and 6 Month Follow up Visit
Description: PGIC - score range = 1 - 7. "1" corresponds to "very much improved" and "7" indicates "very much worse" pertaining to overall activity, symptoms, emotions, and quality of life. The means of these scores and their respective standard deviations are reported for each study group.
Time Frame: Baseline and 6 months
Population: Six subjects in the TransDiscal System study arm, and seven subjects in the Medical Management study arm did not provide follow-up data.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | TransDiscal System | Medical Management
Number analyzed (Participants) | 23 | 27
units on a scale | -1.7 (1.6) | 0.3 (1.5)

7. Secondary Outcome: Mean Change in Score of Oswestry Disability Index (ODI) Between Screening and 6 Month Follow up Visit
Description: ODI - score range = 0 - 100. "0" corresponds to "no disability" and "100" indicates the "maximum disability possible". The means of these scores and their respective standard deviations are reported for each study group.
Time Frame: Baseline and 6 Months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TransDiscal System | Medical Management
Number analyzed (Participants) | 24 | 27
units on a scale | -11 (17) | 0.22 (7)

ADVERSE EVENTS:
Arm/Group | TransDiscal System | Medical Management
Serious Adverse Events (participants affected / at risk) | 3/29 | 1/34
Other Adverse Events (participants affected / at risk) | 24/29 | 23/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TransDiscal System (N=29) | Medical Management (N=34)
pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
chest pain (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TransDiscal System (N=29) | Medical Management (N=34)
vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
discomfort (General disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 1 (1) | 0 (0)
inflammation (General disorders) | 0 (0) | 1 (1)
pain (General disorders) | 3 (3) | 3 (3)
swelling (General disorders) | 0 (0) | 1 (1)
seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
sinusitis (Infections and infestations) | 0 (0) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
influenza (Infections and infestations) | 1 (1) | 0 (0)
foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 9 (9)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
bunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 1 (1) | 1 (1)
migraine (Nervous system disorders) | 0 (0) | 1 (1)
dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
parathesia (Nervous system disorders) | 2 (2) | 1 (1)
sciatica (Nervous system disorders) | 1 (1) | 1 (1)
depression (Psychiatric disorders) | 2 (2) | 1 (1)
insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
loss of bladder sensation (Renal and urinary disorders) | 0 (0) | 1 (1)
pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No